CLINICAL TRIAL: NCT05235230
Title: A Randomized, Single-dose, Partial Replicate, Three-phase, Three-sequence, Open-label, Bioequivalence Study Comparing Quetiapine 25 mg in Different Products After Oral Administration to Healthy Adult Subjects Under Fasting Conditions
Brief Title: Partially Replicate Bioequivalence Study of Quetiapine 25 mg in Healthy Volunteers Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Hala Masoud, FRC Technical Director & CEO, Future University in Egypt
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: QUE-B-21-045
Record Dates: First submitted 2022-01-31; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Bioequivalence
Keywords: Quetiapine; Replicate; Randomized

STUDY DESIGN:
Intervention Model Description: A randomized, single-dose, partial replicate crossover, three-phase, three-sequence, two treatments bioequivalence study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product (T) 25 mg Film Coated Tablets (Experimental): Single oral dose of 25 mg tablet
  Interventions: Drug: Test product (T) 25 mg Film Coated Tablets
- Reference product (R) 25 mg Film Coated Tablets (first dose) (Active Comparator): Single oral dose of 25 mg tablet
  Interventions: Drug: Reference product (R) 25 mg Film Coated Tablets
- Reference product (R) 25 mg Film Coated Tablets (second dose) (Active Comparator): Single oral dose of 25 mg tablet
  Interventions: Drug: Reference product (R) 25 mg Film Coated Tablets

INTERVENTIONS:
Drug: Test product (T) 25 mg Film Coated Tablets — Film Coated Tablets products containing 25 mg Quetiapine
  Arms: Test product (T) 25 mg Film Coated Tablets
Drug: Reference product (R) 25 mg Film Coated Tablets — Reference product (R) 25 mg Film Coated Tablets
  Arms: Reference product (R) 25 mg Film Coated Tablets (first dose); Reference product (R) 25 mg Film Coated Tablets (second dose)

SUMMARY:
The current study is conducted to evaluate and compare the relative bioavailability for Quetiapine in two different products containing 25 mg Quetiapine after a single oral dose administration under fasting conditions.

DETAILED DESCRIPTION:
A randomized, single-dose, partial replicate, three-phase, three-sequence, bioequivalence study of the two study products. Blood samples were collected at different time intervals and stored at -70⁰C freezer. Quetiapine plasma concentrations were analyzed using a validated LC-MS-MS method then pharmacokinetics and statistical analysis were performed on the concentrations obtained using Phoenix WinNonlin® software.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained for study.
* Age 18 - 55 years,
* Body mass index between 18.5 and 30 kg/m2
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination.
* Vital signs without significant deviations.
* All laboratory screening results are within the normal range or clinically non-significant.

Exclusion Criteria:

* History or presence of any disorder or condition that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the investigator.
* History of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, allergic, dermatologic, hematologic, neurologic, or psychiatric disease, or cancer.
* Any confirmed significant allergic reactions against any drug, or multiple allergies.
* Clinically significant illness 28 days before study phase I.
* Alcohol or any solvent intake.
* Regular use of medication.
* Positive urine screening of drugs of abuse.
* Use of any systemic medications (prescription medications, OTC products, supplements, or herbal preparations) for 14 days prior to dosing and during the study.
* History or presence of significant smoking (more than one pack per day cigarettes) or refusal to abstain from smoking for 48 hours before dosing until checkout.
* Blood donation within the past 60 days.
* Participation in another bioequivalence study within 60 days prior to the start of phase I of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Pre-dose (0), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12 and 24 hours post dose
  Cmax is observed as the maximum of Quetiapine peak concentration
Area under the plasma concentration curve from administration to last observed concentration at time t (AUC(0-t)) | Pre-dose (0), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12 and 24 hours post dose
  The AUC (0-t) is the area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (tlast)
Area under the plasma concentration curve extrapolated to infinite time (AUC(0-inf)) | Pre-dose (0), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12 and 24 hours post dose
  AUC(0-inf) "the area under the curve," which is a way of measuring the total amount of the active drug in a subject's system over a period of time from administration ("0") to the time that the drug is no longer present in the subject's body ("infinity")

SECONDARY OUTCOMES:
Maximum time (Tmax) | Pre-dose (0), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12 and 24 hours post dose
  Time until Cmax is reached
Elimination Rate Constant (Kel) | Pre-dose (0), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12 and 24 hours post dose
  Kel is a value used in pharmacokinetics to describe the rate at which a drug is removed from the human system
Plasma concentration half-life (t1/2) | Pre-dose (0), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12 and 24 hours post dose
  t1/2 is the time taken for the plasma concentration of a drug to reduce to half its original value. It is used to estimate how long it takes for a drug to be removed from your body.

CONTACTS AND LOCATIONS:
Locations (1):
- Future Research Center (FRC), Cairo, Egypt